CLINICAL TRIAL: NCT07300813
Title: Clinical Evaluation of Hair Loss, Hair Growth, and Skin Improvement in Human Volunteers Following a Double-blind, Placebo-controlled, 1:1 Randomized Trial of 'Olistic Next Women'
Brief Title: Olistic_2025 for Hair Loss, Hair Growth, and Skin Improvement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bionos Biotech S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Olistic_2025
Record Dates: First submitted 2025-12-04; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hair Care; Hair Loss; Female Pattern Hair Loss
Keywords: Hair density; Female pattern hair loss; Hair growth; Skin aging; Facial wrinkles; Oral nutraceutical; Skin firmness; Skin elasticity; Dietary supplement; Collagen peptides
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to receive either Olistic Next Women or a matching placebo and remain in the same group for the full 6-month treatment period (parallel two-arm design, no crossover).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blind with matching placebo. Participants, care providers, investigators, and outcomes assessors are unaware of treatment allocation. Active product and placebo are identical in appearance, packaging, labeling, and administration schedule. Randomization codes are held by an independent party and will not be broken until database lock, except in case of medical emergency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olistic Next Women (Experimental): This group will be provided with the product Olistic Next Women.
  Interventions: Other: Olistic Next Women
- Placebo (Placebo Comparator): This group will be provided with placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Olistic Next Women — Participants will be provided with Olistic Next Women and instructed to drink one vial orally once daily for 6 months (28 consecutive days followed by 2 days of rest each month). Efficacy will be evaluated at baseline and at approximately 1, 3, and 6 months using HairMetrix® imaging (hair density and growth parameters), standardized hair shedding tests, 3D facial wrinkle imaging, Glossymeter® (shine/brightness), Corneometer® (hydration), Cutometer® (firmness, elasticity, fatigue), and patient-reported questionnaires (Skindex-29 and a self-perception questionnaire). Product is supplied in individual single-dose vials and stored according to the manufacturer's instructions. All procedures occur at Bionos Biotech S.L. facilities.
  Arms: Olistic Next Women
Other: Placebo — Participants will be provided with a matching placebo and instructed to drink one vial orally once daily for 6 months (28 consecutive days followed by 2 days of rest each month). Efficacy will be evaluated at baseline and at approximately 1, 3, and 6 months using HairMetrix® imaging (hair density and growth parameters), standardized hair shedding tests, 3D facial wrinkle imaging, Glossymeter® (shine/brightness), Corneometer® (hydration), Cutometer® (firmness, elasticity, fatigue), and patient-reported questionnaires (Skindex-29 and a self-perception questionnaire). Product is supplied in individual single-dose vials and stored according to the manufacturer's instructions. All procedures occur at Bionos Biotech S.L. facilities.
  Arms: Placebo

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled clinical trial is to find out whether daily oral intake of the nutraceutical Olistic Next Women can reduce hair loss, improve hair growth and quality, and improve signs of skin aging in women with early female-pattern hair loss. One hundred healthy women aged 50-65 years with initial FPHL will be randomly assigned 1:1 to receive either Olistic Next Women or a matching placebo for 6 months. Participants will drink one vial per day for 28 days, rest 2 days each month, and repeat this cycle for the duration of the study.

The main questions are whether Olistic Next Women, compared with placebo, (1) increases hair density and thickness, improves hair growth (anagen/telogen and terminal/vellus ratios), and reduces hair shedding; and (2) improves facial skin parameters related to aging, such as wrinkles, hydration, brightness, elasticity, and firmness. At baseline and at approximately 1, 3, and 6 months, participants will attend clinic visits where hair metrics at two scalp sites will be quantified using HairMetrix imaging; hair shedding will be assessed with standardized comb and wash tests; and hair fiber damage (in a subset) will be evaluated by scanning electron microscopy. Facial skin will be evaluated using 3D wrinkle imaging, Glossymeter, Corneometer, and Cutometer measurements. Participants will also complete the Skindex-29 and a self-perception questionnaire at several time points while maintaining their usual diet and cosmetic routines and avoiding other hair-active treatments or supplements.

DETAILED DESCRIPTION:
Hair loss in women and skin aging are multifactorial processes influenced by intrinsic factors (genetics, hormonal changes, chronological aging) and extrinsic factors (UV exposure, environmental stressors, lifestyle). Female pattern hair loss (FPHL) is characterized by gradual thinning and a reduction in hair density, often associated with a decrease in the terminal/vellus hair ratio and changes in the anagen/telogen balance. In parallel, skin aging manifests as wrinkles, loss of elasticity and firmness, reduced hydration, and altered barrier function. Nutraceuticals containing bioactive compounds such as collagen-derived amino acids, plant extracts, vitamins, and minerals have been proposed as a supportive strategy to improve hair and skin parameters from within.

In this double-blind, placebo-controlled, 1:1 randomized cosmetic study, investigators will assess the efficacy of the oral supplement "Olistic Next Women" on hair loss/growth and age-related skin parameters in healthy adult women with initial FPHL. One hundred volunteers aged 50-65 years with early FPHL, confirmed through dermatological assessment, will be enrolled at Bionos Biotech S.L. (Valencia, Spain) after providing written informed consent and meeting predefined inclusion and exclusion criteria. Participants will be randomized to receive either Olistic Next Women or a matching placebo and will consume one vial daily for 28 consecutive days followed by 2 days of rest each month, for a total treatment duration of 6 months. The product and placebo are manufactured in compliance with relevant EU regulations regarding safety, microbiology, allergens, and heavy metals.

Hair and skin assessments will be performed at baseline and during follow-up visits to enable comparisons over time between active and placebo groups. A dermatologist will conduct an initial hair evaluation, followed by standardized measurements at multiple time points. At baseline (D0), month 3 (D90), and month 6 (D180), hair density and growth parameters will be quantified at two scalp sites (behind the ear and at the top of the head, where FPHL is more evident) using HairMetrix® imaging. Parameters will include terminal/vellus ratio, average hairs per follicular unit, hair width, follicle count per cm², hair count per cm², anagen/telogen ratio, and short-term growth rate. Hair shedding will be evaluated at several visits using standardized comb and wash tests after controlled intervals without washing or combing. In a subset of 10 volunteers, hair fiber damage and integrity will be assessed by scanning electron microscopy. Hair volume, general appearance, and overall hair quality will be graded by clinical scoring, and hair shine will be measured using a Glossymeter® probe.

Facial skin will be evaluated at baseline and follow-up visits using non-invasive instrumental methods. Wrinkle area, depth, and volume will be quantified by 3D imaging; skin brightness will be measured with a Glossymeter®; hydration will be assessed using a Corneometer®; and elasticity and firmness will be measured with a Cutometer®. Participants will also complete the Skindex-29 questionnaire to capture the impact of hair and skin status on quality of life, as well as a self-perception questionnaire to document subjective impressions of hair and skin changes over the course of treatment.

Throughout the study, participants will be instructed to maintain their usual diet and basic hygiene habits, to avoid initiating new oral supplements or systemic/topical products with similar effects to the investigational product, and to refrain from intense or invasive cosmetic treatments. Major changes in hairstyle or routine that could interfere with measurements will not be permitted. Compliance with product intake and study instructions will be supported through written guidelines and regular contact with the research team. The primary analysis will compare changes from baseline to post-treatment time points between the Olistic Next Women and placebo groups using appropriate statistical methods for continuous outcomes, with two-sided tests and a significance level of 0.05. The planned sample size of 100 women is based on prior experience and is expected to provide adequate power to detect clinically relevant differences in key hair and skin parameters.

The study will be conducted in accordance with the Declaration of Helsinki, applicable regulations, and local ethics committee approval. All participants will provide written informed consent prior to any study procedures. Data will be coded and handled under Spanish data protection law, and study records will be retained according to regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with initial FPHL.
* Commitment not to use systemic, topical, or oral products with an effect similar to that of the product to be evaluated throughout the study period.
* Do not change the daily routine regarding the use of cosmetic products and eating habits.
* Commitment to comply with all protocol requirements specified in the subject information sheet.
* Availability to comply with all study visits.

Exclusion Criteria:

* Allergy or reactivity to some of the components of the product, or a product with similar category than tested one.
* Women who have undergone dermatological treatment for hair loss (PRPs, mesotherapy, etc.) or hair transplant.
* Scalp diseases: cicatricial alopecia, alopecia areata, folliculitis decalvans, psoriasis, moderate severe seborrheic dermatitis, eczema, cancer, etc.
* Women who present alopecia because of a medical illness (hypothyroidism, anemia, lupus, etc.).
* Relevant cutaneous marks in the experimental areas, which could interfere with the measurements (scars, sunburns, etc.).
* In-use relevant pharmacological or hormonal treatment (eg. valproic acid, carbamazepine, phenytoin).
* Women with thyroid alteration (hyper- or hypothyroidism)
* Women who have previously participated in similar studies or who have used anti-hair loss products in the last 3 months.
* Women who are being treated with anticoagulants, antifungals, anxiolytics, amphetamines, retinoids, iron, antithyroid, anticonvulsants, beta blockers and/or ACE inhibitors, minoxidil, finasteride, etc.
* Women who started hormonal treatment (oral or topical contraceptives) in the 6 months prior to the start of the study.
* Women who started taking any drug chronically less than 6 months before the start of the study (they should have a stable situation with the medication over 6 months).
* Modification of the usual diet: low-calorie diet, Atkins diet, etc.
* Pregnant, postpartum (6 months) or breastfeeding women, or who intend to get pregnant during the duration of the study.
* Evidence of systemic diseases (e.g. cardiac disease, psychiatric disease, etc.) or gastrointestinal diseases.
* Serious conditions or illnesses that, in the opinion of the researcher, may be aggravated by participation in the study or that put the development of the study at risk.
* Planned hairstyle changes throughout the study
* Presence of skin diseases or melanomas
* Forecast of change of routine or relevant way of life, during the period of study.
* Other exclusion criteria to be added by the customer.
* Women who have gone dermatological treatment, that they have introduced minoxidil (oral or topical) at least 6 months prior, and antiandrogens (e.g. finasteride) at least 12 months before the start of the study.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only participants who self-identify as women are eligible for this study.
Enrollment: 100 (Actual)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in hair density (hair count per cm²) measured by HairMetrix®. | Baseline ( 2 days after clipping) 3 months (2 days after clipping), 6 months (2 days after clipping).
  Change in hair density, expressed as hair count per cm², from baseline to follow-up visits. Hair density is assessed using standardized HairMetrix® imaging at predefined scalp sites. To ensure measurement accuracy and reproducibility, all assessments are performed 2 days after standardized scalp clipping, allowing sufficient hair regrowth for reliable detection and analysis.

SECONDARY OUTCOMES:
Change from baseline in terminal/vellus hair ratio (unitless) measured by HairMetrix® | Baseline ( 2 days after clipping) 3 months (2 days after clipping), 6 months (2 days after clipping).
  Change in the terminal-to-vellus hair ratio from baseline to follow-up visits, assessed using standardized HairMetrix® imaging at predefined scalp sites. Measurements are performed 2 days after standardized scalp clipping at each time point to ensure consistent hair length and reliable classification of terminal and vellus hairs.
Change from baseline in mean hair shaft width (µm) measured by HairMetrix® | Baseline ( 2 days after clipping) 3 months (2 days after clipping), 6 months (2 days after clipping).
  Change in mean hair shaft width from baseline to follow-up visits at the predefined scalp site(s). To ensure measurement accuracy and reproducibility, all assessments are performed 2 days after standardized scalp clipping, allowing sufficient hair regrowth for reliable detection and analysis.
Change from baseline in follicle count per cm² measured by HairMetrix® | Baseline ( 2 days after clipping) 3 months (2 days after clipping), 6 months (2 days after clipping).
  Change in follicle count per cm² from baseline to follow-up visits at the predefined scalp site(s). To ensure measurement accuracy and reproducibility, all assessments are performed 2 days after standardized scalp clipping, allowing sufficient hair regrowth for reliable detection and analysis.
Change from baseline in anagen/telogen ratio (unitless) measured by HairMetrix® | Baseline ( 2 days after clipping) 3 months (2 days after clipping), 6 months (2 days after clipping).
  Change in anagen/telogen ratio from baseline to follow-up visits at the predefined scalp site(s). To ensure measurement accuracy and reproducibility, all assessments are performed 2 days after standardized scalp clipping, allowing sufficient hair regrowth for reliable detection and analysis.
Change from baseline in short-term hair growth rate (mm/day) measured by HairMetrix® | Baseline ( 2 days after clipping) 3 months (2 days after clipping), 6 months (2 days after clipping).
  Change in short-term growth rate from baseline to follow-up visits at the predefined scalp site(s). To ensure measurement accuracy and reproducibility, all assessments are performed 2 days after standardized scalp clipping, allowing sufficient hair regrowth for reliable detection and analysis.
Change from baseline in wrinkle volume (mm³) measured by 3D imaging. | Baseline and ~1, 3, 6 months.
  Change in wrinkle volume, expressed in mm³, from baseline to follow-up visits, assessed using standardized VISIA-PRIMOS® 5 three-dimensional facial imaging at predefined facial regions. Image acquisition and analysis are performed under controlled conditions to ensure reproducibility across time points.
Change from baseline in wrinkle area (mm³) measured by 3D imaging | Baseline and ~1, 3, 6 months.
  Change in wrinkle area, expressed in mm³, from baseline to follow-up visits, assessed using standardized VISIA-PRIMOS® 5 three-dimensional facial imaging at predefined facial regions. Image acquisition and analysis are performed under controlled conditions to ensure reproducibility across time points.
Change from baseline in depth volume (mm³) measured by 3D imaging | Baseline and ~1, 3, 6 months.
  Change in wrinkle depth, expressed in mm³, from baseline to follow-up visits, assessed using standardized VISIA-PRIMOS® 5 three-dimensional facial imaging at predefined facial regions. Image acquisition and analysis are performed under controlled conditions to ensure reproducibility across time points.
Change from baseline in skin hydration (Corneometer units, a.u.) | Baseline and ~1, 3, 6 months.
  Change in Corneometer® readings (arbitrary units) from baseline to follow-up visits at the predefined facial region(s).
Change from baseline in skin gloss/brightness (Gloss units) | Baseline and ~1, 3, 6 months.
  Change in Glossymeter® readings from baseline to follow-up visits at the predefined facial region(s).
Change from baseline in skin elasticity (Cutometer® R2, unitless) | Baseline and ~1, 3, 6 months.
  Change in skin elasticity, expressed by the R2 parameter (mm), from baseline to follow-up visits. Measurements are performed using a Cutometer® at predefined facial regions under standardized conditions to ensure reproducibility across all time points.
Change from baseline in skin firmness (Cutometer® R0, mm) | Baseline and ~1, 3, 6 months.
  Change in skin firmness, expressed by the R0 parameter (mm), from baseline to follow-up visits. Measurements are performed using a Cutometer® at predefined facial regions under standardized conditions to ensure reproducibility across all time points.
Change from baseline in Skindex-29 overall score (0-100; higher = worse quality of life) | before treatment, after 1-, 3 and 6 months treatment.
  Change in the total score of the Skindex-29 questionnaire from baseline to follow-up visits. The Skindex-29 is a 29-item, patient-reported questionnaire assessing the impact of alopecia and scalp-related symptoms on quality of life (e.g., pain, itching, burning, irritation, emotional distress, social functioning, daily activities, and sexual life). Each item is scored on a 5-point Likert scale ranging from 0 (Never) to 4 (All the time). The total score ranges from 0 to 116, with higher scores indicating worse quality of life.
Change from baseline in Self-Perception Questionnaire total score | before treatment, after 1-, 3 and 6 months treatment.
  Change in participants' self-assessment of product performance and cosmetic acceptability from baseline to follow-up visits. Each parameter is rated on a 5-point agreement scale ranging from 1 (Agree), 2 (Partially agree), 3 (Slightly agree), 4 (Partially disagree) to 5 (Disagree).
  For data analysis, an overall acceptance score is calculated as the percentage of positive evaluations (responses of Agree, Partially agree, or Slightly agree) across all assessed parameters. An overall acceptance value ≥ 80% is considered indicative of high consumer acceptance.
Change from baseline in hair volume, general appearance, and hair quality assessed by clinical scoring | Baseline and ~1, 3, 6 months.
  Change in hair volume, general appearance, and overall hair quality from baseline to follow-up visits, assessed using standardized clinical scoring. Evaluations are performed at predefined time points based on standardized photographs. Images are independently analyzed by external dermatologists blinded to treatment allocation to ensure objective assessment.
Change from baseline in hair fiber integrity and thickness assessed by scanning electron microscopy | Baseline and ~1, 3, 6 months.
  Change in hair fiber integrity and thickness from baseline to follow-up visits, assessed using scanning electron microscopy (SEM) in a subset of 10 volunteers. SEM imaging is used to evaluate hair fiber surface morphology and structural damage, allowing qualitative and semi-quantitative assessment of fiber integrity and thickness over time.
Change from baseline in number of fallen hairs after combing assessed by comb test | Baseline and ~1, 3, 6 months.
  Change in the number of fallen hairs collected after standardized combing from baseline to follow-up visits, assessed using a comb test procedure. This outcome is used to evaluate changes in hair shedding and to assess a potential strengthening effect over time.
Change from baseline in number of fallen hairs after washing assessed by wash test | Baseline and ~1, 3, 6 months.
  Change in the number of fallen hairs collected after a standardized washing procedure from baseline to follow-up visits, assessed using a wash test procedure. This outcome is used to evaluate changes in hair shedding and to assess a potential strengthening effect over time.

CONTACTS AND LOCATIONS:
Overall Officials: Adela Serrano Gimeno, PhD, Principal Investigator — Bionos Biotech S.L. , LabAnalysis Life Science
Locations (1):
- Bionos Biotech S.L., LabAnalysis Life Science, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No